CLINICAL TRIAL: NCT02880566
Title: Efficacy of Scalp Block on Hemodynamic Stability and Opioid Consumption During Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor and Chair, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: anesneuro2016001
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Craniotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Full scalp block performed with a total of 30 ml of levobupivacaine 0.33 %.
  Interventions: Procedure: Scalp block
- Control (Placebo Comparator): Full scalp block performed with a total of 30 ml of normal saline.
  Interventions: Procedure: Scalp block

INTERVENTIONS:
Procedure: Scalp block — Full scalp block

SUMMARY:
Prospective randomised double-blinded placebo-controlled trial on the efficacy of scalp blocks on hemodynamic stability and opioid consumption during and after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective craniotomy for supratentorial lesion

Exclusion Criteria:

* Allergy to local anaesthetic
* Psychiatric disease
* Inability to consent
* Uncontrolled intracranial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic stability | 5 minutes
  Increased in mean arterial pressure or heart rate of more than 15 % within 5 minutes of head pinning

SECONDARY OUTCOMES:
Cumulative intraoperative remifentanil consumption | 24 hours
Cumulative postoperative morphine consumption | 48 hours
Postoperative pain scores | 48 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carella M, Tran G, Bonhomme VL, Franssen C. Influence of Levobupivacaine Regional Scalp Block on Hemodynamic Stability, Intra- and Postoperative Opioid Consumption in Supratentorial Craniotomies: A Randomized Controlled Trial. Anesth Analg. 2021 Feb 1;132(2):500-511. doi: 10.1213/ANE.0000000000005230. PMID 33060491